CLINICAL TRIAL: NCT03428555
Title: Is an Integrated Care Pathway for Adolescents With Depression More Effective Than Treatment as Usual? A Controlled Clinical Trial
Brief Title: Integrated Care Pathway for Youth Depression
Acronym: CARIBOU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Darren Courtney, Principle Investigator, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 079/2017
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: ICP1; Depression; Adolescent Behavior
MeSH Terms: conditions — Depression; Adolescent Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Intervention Arm (n=30 over 17 months at, CAMH): The intervention is an integrated care pathway and Comparison Arm- Treatment As Usual (n=30 over 17 months at SHSC):
Masking Description: Participants are not blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrate Care Pathway (Experimental): The intervention is an Integrated Care Pathway with 3 key components.
  1. Clinical Practice Guidelines (CPG) recommendations: The initial template of the treatment protocol was based on the NICE CPGs for Depression in Children and Young People.
  2. Provider engagement: The clinicians at CAMH reviewed the template and collaboratively developed a flow chart defining the treatment protocol.
  3. Measurement-based care: Feedback measures are taken every four weeks and the results are provided to the clinician, patient and family to inform treatment decisions. The feedback measures are the Mood and Feelings Questionnaire, the Columbia Impairment Scale (CIS) and the General Functioning Domain of the McMaster Family Assessment Device (MFAD).
  Interventions: Behavioral: Integrated Care Pathway
- Treatment As Usual (Active Comparator): Treatment As Usual : Participants at SHSC will receive treatment at could include a psychiatric evaluation, possible medication management and various types of psychotherapy, including cognitive-behavioural therapy, interpersonal psychotherapy, psychodynamic psychotherapy and family therapy. There is no structured protocol and no systematic Measurement Based Care. A research assistant will record the interventions received in either group via chart review.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Integrated Care Pathway — The intervention is a integrated care pathway based on the NICE Clinical Practice Guidelines and measurement-based care in the form of a flow chart. Each decision point on the pathway is guided by results of self-report measures for depression (the Mood and Feelings Questionnaire), functional impairment (Columbia Impairment Scales) and family functioning (the McMaster Family Assessment Device). The results of these scales and protocol recommendations are fed back to the patients, families and clinicians in order to make further treatment decisions
  Arms: Integrate Care Pathway
Behavioral: Treatment As Usual — Treatment As Usual represents what clinicians would typically do when presented with an adolescent with depression. There is no algorithm provided to guide clinical decision-making and no systematic measurement-based care.
  Arms: Treatment As Usual

SUMMARY:
Major Depressive Disorder in adolescence is prevalent and debilitating. Our group aims to improve treatment response through the use of an Integrated Care Pathway (ICP) based on a high quality Clinical Practice Guideline and measurement-based care (MBC; where periodic symptom scale scores are used to make treatment decisions). We propose a controlled clinical trial comparing ICP to treatment-as-usual (TAU) across two sites.

DETAILED DESCRIPTION:
Background: There is a gap between what is known from the evidence about the treatment of adolescent depression and what is practiced. Moreover, while there is evidence that measurement-based care can improve outcomes for adults with various mental health conditions, there is limited information on this framework in adolescent depression.

Objective: Our study aims to enhance the implementation of evidence-based care (using the NICE Clinical Practice Guidelines as a template) combined wtih measurement-based care through the use of an Integrated Care Pathway (ICP) in adolescents with depression.

Hypothesis: As this is a pilot study, our hypotheses centre around feasibility. We hypothesize that: (1) we will recruit at least 30 participants to the ICP treatment arm and 30 participants at the "treatment-as-usual" arm at a different site (2) that baseline measures will be fully completed by 95% of adolescents recruited, (3) that baseline measures will take 2 hours to complete for adolescents and 1 hour to complete for caregivers, (4) that a mean of 90% of the key aspects of the treatment protocol are followed in the ICP group (5) that 80% of participants recruited will complete measures at the end of the 20-week interval and that (6) 90% of the youth, caregivers and clinicians who partake int eh study will attend a focus group to provide qualitative feedback on their experience.

Design: This is a non-randomized controlled clinical trial. Randomizing at the individual level is not possible - the intervention is implemented at the clinic level; so the effect of the intervention on one youth within a clinic would influence the care of other youth at the clinic.

Sampling: Participants are recruited from psychiatric clinics at 2 sites. Each site will recruit to their respective treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatrist's impression is that depression is a primary psychiatric. concern
* 14-18 years old.
* DSM-5 criteria for Major Depressive Disorder or Persistent Depressive Disorder as per the Diagnostic Interview for Affective Symptoms for Children (DIAS-C19).
* Speak, read and write English at a grade 6 level.

Exclusion Criteria:

* Threshold psychotic symptoms.
* Bipolar disorder.
* Moderate-to-severe substance use disorder.
* Autistic spectrum disorder or intellectual disability.
* Eating disorder.
* Suicide-related behaviours requiring acute intervention.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-08-29 (Estimated); Study Completion 2020-02-21 (Estimated)

PRIMARY OUTCOMES:
Change in Childhood Depression Rating Scale-Revised scores | 20 weeks
  The CDRS-R is a 17-item measure rated by an evaluator after a semi-structured interview with the adolescent relating to symptoms of depression over the past 2 weeks. Scores range from 0 to 100 with a score of over 55 interpreted as a moderate to severe rating. Lower values represent a better outcome.

SECONDARY OUTCOMES:
Change in WHO Disability Assessment Schedule 2.0 for Children And Youth | 20 weeks
  Change in function as reported by participant The sum of scores of the items across all domains constitutes a statistic that is sufficient to describe the degree of functional limitations. Lower values represent a decrease in their subjective depression rating over the previous 2 weeks.
Change in Childhood Behaviour Checklist | 20 weeks
  Change in overall psychopathology as reported by caregiver.Total scores may be computed for Social Competence, Behavior Problems, Internalizing Problems, and Externalizing Problems, plus scores for each of the 8 syndrome scales. Raw scores are converted to age-standardized scores (T-Scores). T scores less than 67 are considered in the normal range, T scores ranging from 67-70 are considered to be borderline clinical, and T scores above 70 are in the clinical range.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szatmari, MD, Study Director — The Center for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - The Center for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- [Derived] Courtney DB, Cheung A, Henderson J, Bennett K, Wang W, Chen S, Battaglia M, Strauss J, Mitchell R, Wang K, Relihan J, Prebeg M, Darnay K, Szatmari P. CARIBOU-1: A pilot controlled trial of an Integrated Care Pathway for the treatment of depression in adolescents. JCPP Adv. 2022 May 27;2(2):e12083. doi: 10.1002/jcv2.12083. eCollection 2022 Jun. PMID 37431464